CLINICAL TRIAL: NCT06732154
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Injection of HRS-5632 in Healthy Subjects - A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study
Brief Title: A Phase I Clinical Study of a Single Subcutaneous Injection of HRS-5632 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5632-101
Record Dates: First submitted 2024-11-12; First posted 2024-12-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-5632 (Experimental)
  Interventions: Drug: HRS-5632
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-5632 — HRS-5632 Injection
  Arms: HRS-5632
Drug: Placebo — Sodium chloride injection
  Arms: Placebo

SUMMARY:
The study is being conducted to evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of HRS-5632 Following a Single Subcutaneous Injection in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Understand the specific procedures of the trial, voluntarily participate in this trial, and sign an informed consent form;
2. Age on the day of signing the informed consent form must be ≥18 and ≤55 years old (inclusive of boundary values);
3. Male subjects must weigh ≥50 kg and female subjects must weigh ≥45 kg, with a Body Mass Index (BMI) within the range of 19 to 30 kg/m² (inclusive of boundary values);
4. Female subjects with childbearing potential must agree to use effective contraception and avoid donating eggs from the time of signing the informed consent form until the end of the trial. Serum pregnancy tests within 7 days before the first dosing and during the trial must be negative, and they must not be breastfeeding; Male subjects with partners who have childbearing potential must agree to use effective contraception and avoid donating sperm from the time of signing the informed consent form until 6 months after the last administration of the trial medication;
5. Vital signs, physical examinations, and laboratory tests (complete blood count, urinalysis, blood biochemistry, coagulation function, thyroid function, sex hormones), 12-lead electrocardiogram, chest X-ray, and abdominal ultrasound must be normal or have abnormalities without clinical significance.

Exclusion Criteria:

1. Subjects with any clinically significant diseases or medical history in the circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric, and metabolic systems, or any other diseases or histories that could interfere with the trial results or any significant laboratory abnormalities judged by the investigator to be clinically meaningful;
2. History of malignant tumors;
3. Use of any prescription, over-the-counter, or traditional Chinese medicine within 14 days prior to the study drug administration, or within 7 half-lives of the drug at the time of screening;
4. Participation in any clinical trial of drugs or medical devices within the last 3 months, or still within 7 half-lives of the drug at the time of screening (the longer standard shall prevail if both are met);
5. Subjects who plan to take lipid-lowering or lipid-affecting drugs not part of this study during the trial;
6. Elevated high-sensitivity C-reactive protein >1.5 times the upper limit of normal, or prothrombin time/international normalized ratio (PT/INR), activated partial thromboplastin time (APTT) >1.25 times the upper limit of normal during the screening period;
7. Positive results in infectious disease screening (including hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, human immunodeficiency virus antibody, syphilis spirochete antibody);
8. Abnormal 12-lead electrocardiogram with clinical significance, or electrocardiogram QT interval (QTcF) > 450 ms in males, > 470 ms in females;
9. Blood donation or blood loss of ≥ 200 mL within the last month before dosing, or ≥ 400 mL within the last 3 months before dosing, or receipt of blood transfusion within the last 8 weeks;
10. History of severe infection, severe trauma, or major surgery within the last 3 months before dosing; planning to undergo surgery during the trial and within two weeks after trial completion;
11. Suspected history of allergy to the study drug or any component of the study drug, allergic constitution, or history of severe drug allergies;
12. History of difficulty with blood draws or intolerance to venipuncture, such as fainting at the sight of needles or blood;
13. Glomerular filtration rate (eGFR) below 60 mL/min/1.73 m² (estimated using the CKD-EPI equation);
14. Average daily smoking of ≥ 5 cigarettes in the three months before dosing; average daily alcohol intake exceeding 15 g in the month before dosing (5 g of alcohol is equivalent to 150 mL of beer, 50 mL of wine, about 17 mL of low-proof spirits, or 10 mL of high-proof spirits);
15. Positive drug screen at the screening visit or positive alcohol breath test;
16. For subjects participating in QT/QTc studies:

1) Heart rate >100 bpm, congenital QT interval prolongation syndrome, or family history of congenital QT interval prolongation, with implanted pacemakers, automatic implantable cardioverter-defibrillators; 2) Use of antiarrhythmic drugs, cardiac drugs, beta-blockers, calcium channel blockers, quinolones, and other drugs that prolong QT/QTc interval or cause risk of torsades de pointes (TdP) within 4 weeks before the first use of the trial drug; 17. Any other conditions deemed by the investigator to make the subject unsuitable for participation in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The percentage of all reported adverse events, serious adverse events and treatment-related adverse events, serious adverse events. | from the single dose administration (Day 1) to Day 337

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) of HRS-5632 | Following a single subcutaneous injection（Day1）to Day4,
Maximum observed drug concentration (Cmax) of HRS-5632 | Following a single subcutaneous injection（Day1）to Day4,

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided